CLINICAL TRIAL: NCT00914498
Title: The Effect of Pre-incisional Local Xylocaine Injection on Post Operative Pain and Scar Formation After Cesarean Section
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Baruch Padeh Medical Center, Poriya (Other Government)
Responsible Party: Izhar Ben-Shlomo, MD, Senior Obstetrician & Gynecologist, The Baruch Padeh Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Xylocaine CS Scar.CTIL
Record Dates: First submitted 2009-06-04; First posted 2009-06-05 (Estimated); Last update posted 2009-08-25 (Estimated); Status verified 2009-08

CONDITIONS: Pain Relief
Keywords: Xylocaine; Casarean section; Post operative pain; Scar quality
MeSH Terms: conditions — Pain, Postoperative | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Xylocaine (Experimental): Participants will receive local injection of 20 ml 1% Xylocaine to the skin incision site
  Interventions: Drug: Local, pre-incisional injection of 20 ml 1% xylocaine
- Controls (Placebo Comparator): Participants will receive injection of 0.9% NaCl 20 ml to the incision site
  Interventions: Drug: Local, pre-incisional injection of 20 ml 1% xylocaine

INTERVENTIONS:
Drug: Local, pre-incisional injection of 20 ml 1% xylocaine — Local, pre-incisional injection of 20 ml 1% xylocaine

SUMMARY:
This study will examine whether pre-incision infiltration of the skin cut site can attenuate post operative pain after a cesarean section. One hundred and twenty women will be allocated to get 20 ml of either placebo or 1% xylocaine at the site of skin incision. We will also examine possible effect of this infiltration of parameters of wound heeling and scar formation, six weeks post partum.

DETAILED DESCRIPTION:
Among all other abdominal operations cesarean section is unique in two aspects. First, the requirement for rapid and as painless as possible recovery is not only important for the general good reasons, but there is the newborn baby, who needs maternal care. Second, in many cases the operation recurs in the same site, which may involve higher level of post operative pain.

Application of local anesthetics to the incision site have been tried for abdominal operation in several forms, ranging from pre-incision injection (1-6) through post incision injection (7 ) to indwelling catheter for protracted instillation (8-9). Where tried, these methods mostly contributed to the reduction of post operative pain and patients' satisfaction, although there is no consensus as to its efficacy. Yet, local, pre-incision injection of local anesthetics has not been tested for cesarean section.

The above not withstanding, it has been proposed that local infiltration of tissue with xylocaine may interfere with wound healing (10-11). Others suggested possible benefit due to antimicrobial activity (12) Conversely, Al- Asfour et al. (13) found no effect of topical oral application of xylocaine on experimental wounds in rabbits. Interestingly, Drucker et al. found that less collagen was deposited in healing wounds that were infiltrated with xylocaine prior to incision, while the strength of the scar was not affected (14-15).

Our proposed study will examine whether pre-incision infiltration of the skin cut site can attenuate post operative pain after a cesarean section. It will also examine possible effect of this infiltration of parameters of wound heeling and scar formation.

ELIGIBILITY:
Inclusion Criteria:

* Candidates for non-emergency cesarean section

Exclusion Criteria:

* Emergency cesarean section
* Known or suspected sensitivity to local anesthetics
* Pre-eclamptic toxemia
* Deranged liver function
* Deranged hemostasis
* Lack of adequate verbal communication

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Level of post operative pain on a visual analog scale | Up to 48 hours postoperative

SECONDARY OUTCOMES:
Appearance of operative scar, compared to previous scar | 6-8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Izhar Ben-Shlomo, MD, Principal Investigator — Department of Obstetrics & Gynecology, Baruch Padeh Medical Center
Locations (1):
- Department of Obstetrics & Gynecology, Baruch Padeh Medical Center, Poria – Neve Oved, Israel